CLINICAL TRIAL: NCT03928730
Title: Assessment of Ultrasonographic Examination for Maxillofacial Swellings
Brief Title: Evaluation of Oral and Maxillofacial Swellings by Ultrasonographic Features
Acronym: Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarek A Abdelsalam, MD (Other)
Responsible Party: Sponsor-Investigator, Tarek A Abdelsalam, MD, Dentist, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: TAbdallah
Record Dates: First submitted 2019-04-21; First posted 2019-04-26 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Swelling Lips & Face
MeSH Terms: conditions — Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group I (Other): Inflammatory swellings
  Interventions: Procedure: resection and removal
- Group II (Other): Cystic swellings
  Interventions: Procedure: resection and removal
- Group III (Other): Lymph node swellings
  Interventions: Procedure: resection and removal
- Group IV (Other): Benign swellings
  Interventions: Procedure: resection and removal
- Group V (Other): Malignant swellings
  Interventions: Procedure: resection and removal

INTERVENTIONS:
Procedure: resection and removal — Surgical resection or removal for histopathological examination

SUMMARY:
Fifty patients were randomly selected with oral and/or maxillofacial swelling, thorough case history and clinical examination were done, then ultrasound examinations were done for all of them and they were classified into five groups (I. inflammatory/space infection and abscess swellings), (II. cystic swellings), (III. lymph node swellings), (IV. benign swellings) and (V. malignant neoplastic swellings) according to their ultrasound features. The patients were subjected to histopathologic evaluation.

DETAILED DESCRIPTION:
Fifty patients with swellings in the oral and/or maxillofacial region were randomly selected. Any other swellings that were caused by trauma and/or fracture, extended below the neck or patient reluctant to undergo US were excluded from the study. This study was approved by the (Research Ethics Committee) (REC), Faculty of Dentistry, Minia University before starting the research and all the entire patients had signed a standardized informed consent laid down by REC.

A comprehensive questionnaire was used to assess history and through extra-oral & intra-oral examinations were carried out and recorded on the basis of criteria reported by Das.11 The ultrasonographic investigations were carried using an ultrasound diagnostic modality (LOGIQ- P5) (GE Medical System, Korea) with color Doppler function by using a linear array transducer, operating at a frequency of (7.5-12 MHz). All the examinations were performed over the swellings and also compared to the contra-lateral/normal side whenever needed. (Fig. 1) All sonographic images were interpreted by an expert sonologist (15 years experience) and US features were recorded to extract ultrasonographic guided (USG) diagnosis and patient's swellings were categorized into five groups: inflammatory/infection/abscess swellings (Group I), cystic swellings (Group II), lymph node swellings (Group III), benign swellings (Group IV) and malignant neoplastic swellings (Group V).12 Finally, the included patients were subjected to either fine needle aspiration cytology (FNAC) or surgical intervention for histopathological examination to extract the histopathological diagnosis

ELIGIBILITY:
Inclusion Criteria:

* All with oral and/or maxillofacial swelling,

Exclusion Criteria:

* Any other swellings that were caused by trauma and/or fracture, extended below the neck or patient reluctant to undergo US were excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Correlation between ultrasonographic features and swellings types | 2 months
  Correlation between ultrasonographic features and swellings types

CONTACTS AND LOCATIONS:
Locations (1):
- MiniaU, Minya, Egypt